## Human Urinary Kallidinogenase Improve Short Term Motor Functional Outcome By Reducing The Corticospinal Tract Damage In Acute Ischemia Stroke Patients

**Central Contact Person:Peifang Li** 

**Telephone:** +8615203216570

**Department: Department of Neurology** 

Responsible institution: The Second Hospital of Hebei Medical

University

Date: 2019.07.15

## **Statistical Analysis Plan**

- Project name: Human urinary kallidinogenase improve short term motor functional outcome by reducing the corticospinal tract damage in acute ischemia stroke patients
- Purpose: This study aimed to assess the effect of Human urinary kallidinogenase on motor functional outcome and relative corticospinal tract damage recovery in the patients with AIS.
- Statistical analysis: The categorical variables were expressed as frequencies and percentages, and the radios were compared by the  $\chi^2$  or Fisher exact test; continuous variables were expressed as means  $\pm$  standard deviation (SD) and were compared by Student's t test. Non-normally distributed continuous variables were presented as median (interquartile range) and compared between groups using Mann-Whitney U test for independent samples and Wilcoxon test for compared samples. P<0.05 was considered to indicate a statistically significant difference between values. The Spearman bivariate correlation was used to examine relationships between NIHSS, mRS, BI scores at discharge and initial VEGF, MBP concentrations, DTT classification, sex, age, previous stroke, intracranial arterial stenosis, comorbidities, FA values, ADC values. Variables with P 0.1 were entered into the multivariable linear regression with the discharge NIHSS, mRS, BI scores as dependent variable and the intercept set to the origin. The measurement data were analyzed by the SPSS 21.0 statistical analytical software (IBM, Armonk, NY, USA).